CLINICAL TRIAL: NCT07017530
Title: Combined Intervention of Cognitive Training and Supervised Physical Exercise for Women With Breast Cancer and Chemotherapy-Related Cognitive Impairment: Study Protocol for a Randomized Controlled Trial
Brief Title: Cognitive Training and Exercise for Women With Breast Cancer and Cognitive Impairment
Acronym: CHEMO-CogEx
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Noelia Durán, Principal Investigator, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI 044/23
Record Dates: First submitted 2025-05-14; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Chemotherapy-Related Cognitive Impairment; Cognitive Training; Exercise; Oncology Nursing
MeSH Terms: conditions — Breast Neoplasms; Chemotherapy-Related Cognitive Impairment; Motor Activity | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cognitive training + exercise group during chemotherapy (Experimental): Al list two cycles of chemotherapy.
  Interventions: Other: Cognitive training
- Cognitive training + exercise group after chemotherapy (Experimental): Al list six months after the completion of chemotherapy.
  Interventions: Other: Cognitive training
- Psychoeducational therapy during chemotherapy (Active Comparator): Al list two cycles of chemotherapy.
  Interventions: Other: Psychoeducational therapy
- Psychoeducational therapy after chemotherapy (Active Comparator): Al list six months after the completion of chemotherapy.
  Interventions: Other: Psychoeducational therapy

INTERVENTIONS:
Other: Cognitive training — Combined Intervention of Cognitive Training and Supervised Physical Exercise
  Other Names: Adapted physical activity
  Arms: Cognitive training + exercise group after chemotherapy; Cognitive training + exercise group during chemotherapy
Other: Psychoeducational therapy — According to standard clinical practice
  Arms: Psychoeducational therapy after chemotherapy; Psychoeducational therapy during chemotherapy

SUMMARY:
Chemotherapy-related cognitive impairment is a prevalent and distressing condition among breast cancer survivors, adversely affecting memory, attention, and overall cognitive function, thereby diminishing quality of life. Emerging evidence suggests that multimodal interventions combining cognitive training and adapted physical exercise may mitigate these cognitive deficits and associated symptoms. This study aims to evaluate the efficacy of a 12-week structured intervention integrating cognitive training and supervised physical exercise in improving cognitive function, fatigue, sleep quality, psychological distress, and overall well-being in women with breast cancer. Furthermore, it seeks to determine the optimal timing for such interventions to maximize their effectiveness. A randomized controlled trial involving 220 participants will assess subjective and objective cognitive outcomes, brain activity, and physical performance. The findings from this research may contribute to the development of evidence-based rehabilitation strategies, enhancing cognitive health and quality of life in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older who were diagnosed with stage 0 to IV breast cancer.
* Women undergoing chemotherapy (at least two cycles) or having completed it at least six months earlier.
* Cognitive impairment must be reported, with scores below 54 on the FACT-Cog scale

Exclusion Criteria:

* Women with significant neurological conditions.
* Women with psychiatric conditions.
* Women with contraindications for physical exercise.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Subjetive Cognitive function | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be assessed using subjective cognitive function measured by Functional Assessment of Cancer Therapy-Cognition (FACT-Cog) scale.
Objective Cognitive Function | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be assessed with Near Infrared Spectroscopy (regional cerebral oxygen saturation).

SECONDARY OUTCOMES:
Fatigue | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be measured with the Fatigue Symptom Inventory (FSI), which assesses the frequency, severity, and perceived interference of fatigue in daily life over the past week
Sleep quality | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a well-validated questionnaire that evaluates sleep across seven components, including latency, duration, efficiency, disturbances, and the use of sleep medications
Insomnia | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be assessed using the Insomnia Severity Index (ISI). This validated questionnaire consists of seven items that evaluate difficulties with sleep onset, sleep maintenance, and early morning awakening, as well as satisfaction with sleep patterns, interference with daily functioning, perceived impairment, and distress caused by sleep problems
Psychological distress | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  Psychological distress will be assessed using the Hospital Anxiety and Depression Scale (HADS).
  The HADS consists of 14 items, each scored from 0 to 3, yielding subscale scores for anxiety (HADS-A) and depression (HADS-D) that each range from 0 to 21, with higher scores indicating greater psychological distress (worse outcome). The total score ranges from 0 to 42.
Quality of life (QoL) | - Baseline - 12 weeks for intervention group - 16 weeks for control group
  It will be measured using the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30)
Abdominal flexor endurance | - Baseline - 12 weeks for intervention group
  It will be assessed using the McQuade Test (seconds)
Upper body and back muscular strength | - Baseline - 12 weeks for intervention group
  It will be assessed using trunk dynamometry (kg)
Lower body endurance | - Baseline - 12 weeks for intervention group
  It will be assessed using the 30-second sit-to-stand test (number of repetitions). The outcome is the number of repetitions completed, with a higher score indicating better lower limb strength and endurance.
Perceived physical fitness | - Baseline - 12 weeks for intervention group
  It will be assessed using the International Fitness Scale (IFIS). It comprises 5 items that evaluate overall fitness, cardiorespiratory fitness, muscular strength, speed-agility, and flexibility. Each item is rated on a 5-point Likert scale ranging from 1 (very poor) to 5 (very good). Higher scores indicate better perceived physical fitness.
Functional exercise capacity | - Baseline - 12 weeks for intervention group
  It will be assessed using the Six-Minute Walk Test (6MWT) (metres)
Perceived effort | - 12 weeks for intervention group
  It will be assessed using the Borg Scale of Perceived Exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud, Badajoz, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No